CLINICAL TRIAL: NCT07154173
Title: Comprehensive Analysis of Gut Microbiota Signatures in Metastatic Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: MCRCGM-SYSU-2025-01
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Rectal Neoplasms; Colon Neoplasms; Microbiota; Metagenome
Keywords: rectal neoplasms; colon neoplasms; microbiota; metagenomics
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — fecal and tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HC: Healthy individuals without colorectal cancer or other cancers Will provide stool samples Matched by age and gender with cancer groups
  Interventions: Procedure: Biospecimen Collection Procedure
- nmCRC: Participants with colorectal cancer without distant metastasis (M0 stage) Confirmed by imaging studies and/or pathological examination Will provide primary tumor tissue, adjacent normal tissue, and stool samples
  Interventions: Procedure: Biospecimen Collection Procedure
- mCRC: Participants with colorectal cancer with distant metastasis (M1 stage) Confirmed by imaging studies and/or pathological examination Will provide primary tumor tissue, metastatic tumor tissue, adjacent normal tissue, and stool samples
  Interventions: Procedure: Biospecimen Collection Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection Procedure — Collection of fecal samples from healthy volunteers, non-metastatic (M0) and metastatic (M1) colorectal cancer patients. Additionally, collection of tissue samples during surgery from operable patients (M0 and M1) for subsequent research analysis.

SUMMARY:
Colorectal cancer (CRC) is one of the most common and deadly cancers worldwide. About 1 in 4 people with CRC already have cancer spread (metastasis) when first diagnosed, and about half develop spread during their illness. Recent research shows that bacteria living in the gut and even within tumors might play an important role in how cancer spreads.

The goal of this study is to better understand how bacteria might influence the spread of colorectal cancer. The main questions the investigators aim to answer are:

Are there differences in bacteria between people whose cancer has spread and those whose cancer has not spread? Could certain bacteria help predict which cancers might spread?

To answer these questions, the investigators will:

Collect different types of samples from participants:

Tumor tissue Normal tissue near the tumor Tissue from where cancer has spread Stool samples before surgery Study the bacteria in these samples using advanced testing methods Compare bacterial patterns between different groups

People can take part in this study if they:

Are between 18 and 75 years old Have colorectal cancer confirmed by doctors Have not taken antibiotics recently Do not have immune system problems

This research may help us:

Understand why some colorectal cancers spread Find new ways to predict which cancers might spread Develop better treatments for colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Pathologically confirmed colorectal cancer
* Clearly defined clinical staging: including imaging or pathologically confirmed metastatic colorectal cancer (stage M1) and colorectal cancer without distant metastasis (stage M0)
* Expected survival ≥ 3 months
* Voluntary participation and signed informed consent

Exclusion Criteria:

* Use of probiotics, antibiotics, or immunosuppressive agents within 1 month before surgery
* Preoperative complete intestinal obstruction or gastrointestinal perforation
* Intraoperative gastrointestinal perforation or tumor rupture
* Previous history of gastrointestinal surgery (excluding colorectal cancer surgery, appendectomy, and cholecystectomy) or concurrent severe gastrointestinal diseases such as inflammatory bowel disease
* Concurrent active systemic immune or infectious diseases, including severe allergies, rheumatoid arthritis, systemic lupus erythematosus, viral hepatitis, acquired immunodeficiency syndrome, etc.
* Concurrent unhealed primary malignant tumors
* Severe organ dysfunction or failure
* Other conditions deemed unsuitable for this study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients aged 18-75 years with pathologically confirmed colorectal cancer treated at the Sixth Affiliated Hospital of Sun Yat-sen University. Participants will be divided into two main groups: those with peritoneal metastasis (metastasis group) and those without distant metastasis (non-metastasis group). The study population will include both male and female patients who meet all inclusion criteria and none of the exclusion criteria. All participants must have clearly defined clinical staging and be scheduled for surgical treatment, with an expected survival of at least 3 months. Patients with recent use of antibiotics, probiotics, or immunosuppressants, those with intestinal obstruction or perforation, and those with other severe comorbidities will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intestinal Microbiota Diversity Differences Between Colorectal Cancer Patients With and Without Peritoneal Metastasis | Fecal samples collected at patient's first hospital admission; tissue specimens collected during surgery. All specimens analyzed within 6 months after collection.
  Comparison of microbial diversity between metastasis and non-metastasis groups, including alpha diversity (Chao1 index for species richness, Shannon index for species diversity) and beta diversity (Bray-Curtis distance, UniFrac distance). These measurements will evaluate differences in intestinal microbiota composition related to colorectal cancer peritoneal metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wirbel J, Pyl PT, Kartal E, Zych K, Kashani A, Milanese A, Fleck JS, Voigt AY, Palleja A, Ponnudurai R, Sunagawa S, Coelho LP, Schrotz-King P, Vogtmann E, Habermann N, Nimeus E, Thomas AM, Manghi P, Gandini S, Serrano D, Mizutani S, Shiroma H, Shiba S, Shibata T, Yachida S, Yamada T, Waldron L, Naccarati A, Segata N, Sinha R, Ulrich CM, Brenner H, Arumugam M, Bork P, Zeller G. Meta-analysis of fecal metagenomes reveals global microbial signatures that are specific for colorectal cancer. Nat Med. 2019 Apr;25(4):679-689. doi: 10.1038/s41591-019-0406-6. Epub 2019 Apr 1. PMID 30936547